CLINICAL TRIAL: NCT04042636
Title: Epidemiological Patterns for Early Onset and Late Onset Bacteremia After Trauma
Brief Title: Epidemiologic Patterns of Bacteremia After Trauma
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Suk-Kyung, professor, Asan Medical Center
Other Study IDs: AsanMC-Bacteremia
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Bacteremia
Keywords: trauma; CLABSI
MeSH Terms: conditions — Bacteremia; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Patients with Bacteremia after trauma
- 2: Patients with non-bacteremia after trauma

SUMMARY:
Presence of pelvic and liver injury on arrival in ED, gastrointestinal tract perforation and massive transfusion within the first 24 hours after trauma appear a significant risk factor for bacteremia. Scoring with the ISS, intra-abdominal and pelvic injury and presence of transfusion and shock at admission to ED appears a useful tool for identifying trauma patients at increased risk of bacteremia.

DETAILED DESCRIPTION:
Purpose: Bacteremia is a major nosocomial infection problem in view of its high mortality. Bacteremia occurs in trauma patients frequently and increases a morbidity and mortality. The aim of this study was to identify risk factors and to describe epidemiological patterns for early onset (EOB) and late onset (LOB) bacteremia after trauma.

Methods: All trauma patients admitted to surgical intensive care unit (SICU) and general ward (GW) from January 2011 to December 2015 were retrospectively enrolled. The following information was collected for each patient and recorded in a computer database: demography, severity of trauma according to the Injury Severity Score (ISS) and each abbreviated injury score (AIS), severity of coma according to the Glasgow Coma Scale (GCS), presence of shock and transfusion. Early onset bacteremia was defined as EOB when onset occurred within 7 days after trauma, and late onset bacteremia was defined as LOB when appearing after 7 days from trauma.

ELIGIBILITY:
Inclusion Criteria:

* The patients who admitted to intensive care unit (ICU) or general ward (GW) through the emergency department after trauma were studied

Exclusion Criteria:

* Patients who arrived on dead-on arrival

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Asan Medical Center with trauma from January 2011 to December 2015
Sampling Method: Non-Probability Sample
Enrollment: 859 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Risk factor for bacteremia after trauma | 5 years
  finding fisk factor for bacteremia in traumatic patients

SECONDARY OUTCOMES:
Etiology of bacteremia after trauma | 5 years
  distinguishing G(+) cocci, G(-) rod, and candida spp.

CONTACTS AND LOCATIONS:
Locations (1):
- Hakjae Lee, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rello J, Ricart M, Mirelis B, Quintana E, Gurgui M, Net A, Prats G. Nosocomial bacteremia in a medical-surgical intensive care unit: epidemiologic characteristics and factors influencing mortality in 111 episodes. Intensive Care Med. 1994;20(2):94-8. doi: 10.1007/BF01707661. PMID 8201105
- [Result] Antonelli M, Moro ML, D'Errico RR, Conti G, Bufi M, Gasparetto A. Early and late onset bacteremia have different risk factors in trauma patients. Intensive Care Med. 1996 Aug;22(8):735-41. doi: 10.1007/BF01709514. PMID 8880240
- [Result] Menges P, Kessler W, Kloecker C, Feuerherd M, Gaubert S, Diedrich S, van der Linde J, Hegenbart A, Busemann A, Traeger T, Cziupka K, Heidecke CD, Maier S. Surgical trauma and postoperative immune dysfunction. Eur Surg Res. 2012;48(4):180-6. doi: 10.1159/000338196. Epub 2012 May 25. PMID 22653168
- [Result] Niven DJ, Fick GH, Kirkpatrick AW, Grant V, Laupland KB. Cost and outcomes of nosocomial bloodstream infections complicating major traumatic injury. J Hosp Infect. 2010 Dec;76(4):296-9. doi: 10.1016/j.jhin.2010.06.004. Epub 2010 Aug 11. PMID 20705364